CLINICAL TRIAL: NCT06801522
Title: Comparison of the Efficacy of Adrenaline Nasal Pack and Xylometazoline Nasal Drops in Decreasing Nasal Bleeding During Nasotracheal Intubation
Brief Title: Adrenaline Nasal Pack vs Xylometazoline Nasal Drops During Nasotracheal Intubation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shaheed Mohtarma Benazir Bhutto Institue of Trauma (Other)
Responsible Party: Principal Investigator, IQRA ASHRAF, Principal Investigator, Shaheed Mohtarma Benazir Bhutto Institue of Trauma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ERC-000104/SMBBIT/2023
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Nasal Bleeding; Nasotracheal Intubation
Keywords: Nasal bleeding, Nasotracheal intubation, adrenaline pack, xylometazoline nasal drops
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Intervention Model Description: Group Xylometazoline will receive xylometazoline nasal drops and Group Adrenaline will receive adrenaline nasal pack
Who Masked: Outcomes Assessor
Masking Description: This study is single blind, assessor is kept blind because participants are difficult to mask due to well distinguished treatment plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xylometazoline Group (Experimental): Participants in this group will receive xylometazoline nasal drops before nasotracheal intubation
  Interventions: Drug: 0.1% xylometazoline nasal drops
- Adrenaline Group (Active Comparator): Participants in this group will recieve adrenaline nasal packing before nasotracheal intubation
  Interventions: Drug: Adrenaline nasal pack

INTERVENTIONS:
Drug: 0.1% xylometazoline nasal drops — Xylometazoline is direct acting, non selective, adrenergic agonist binding with alpha 1&2 receptors, used for vasoconstriction to decrease nasal bleeding.
  Arms: Xylometazoline Group
Drug: Adrenaline nasal pack — Adrenaline is direct acting, non selective, adrenergic agonist binding with alpha and beta receptors both, used for vasoconstriction to decrease nasal bleeding.
  Arms: Adrenaline Group

SUMMARY:
The goal of this trial is to compare efficacy of xylometazoline nasal drops and adrenaline nasal pack in participants undergoing elective oromaxillofacial surgeries.

The main question aim to answer is xylometazoline nasal drops better than adrenaline nasal packing in terms of nasal bleeding during nasotracheal intubation. Researchers are comparing 2 groups of participants.

Participants in group Xylometazoline are receiving 0.1% xylometaxoline nasal drops.

Participants in group Adrenaline are receiving adrenaline nasal packing.

DETAILED DESCRIPTION:
This study is conducting after permission from institutional ethical committee. Participants came for elective OMF surgery under general anesthesia are enrolled in this study who fulfilled the inclusion criteria. Informed consent is taken from the participants. Brief history about demographic data was taken from each participant. All participants are examined for airway assessment, cardiovascular and respiratory examination before undergoing anesthesia. Participants are divided into 2 groups by simple lottery method in group xylometazoline and group adrenaline.

Group Xylometazoline: receive 3 to 5 drops of 0.1% xylometazoline nasal drops in selected nostril 15 mins before transfer to OT.

Group Adrenaline: receive intranasal packing with adrenaline soaked gauze piece in selected nostril. Packing is done 15 mins before transfer to OT and removed after 7 to 10 minutes. Proper monitoring of vital signs will be done in preoperative area.

Anesthesia machine and accessories are checked, and drugs including emergency drugs are kept ready. Baseline BP, heart rate, ECG, and peripheral oxygen saturation is obtained and recorded from multipara monitor. All participants are preoxygenated by 100% oxygen for 5 mins. Induction is done with propofol (1%) 2mg/kg and atracurium 0.5 mg/kg by senior anesthesiologist present. The anesthetist present in OT is blind to both groups. Laryngoscopy is done by an experienced anesthesiologist using a MAC 3 or 4 blade based on participants' anatomy. Nasotracheal intubation is done by a cuffed lubricated (with lidocaine 2%) nasal tube of appropriate size. Anesthesia is maintained with atracurium 0.1 mg/kg and isoflurane in 60% O2 at 3L flow.

The anesthesiologist will record incidence and severity of bleeding at the time of intubation and extubation.

Data will be analyzed on SPSS version 20. Chi square test will be used to compare the incidence of nasal bleeding in both groups. Effect modifiers are controlled through stratification of age, gender, diabetes mellitus, hypertension to see the effect of these on the outcome variables. Post stratification chi square test will be applied taking P-value of <0.05 as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2
* Age group between 18-60 years
* Mallampati score 1 and 2
* Either gender
* Participants who undergo elective oromaxillofacial surgery

Exclusion Criteria:

* Lack of consent
* Participants with anticipated difficult airway
* Participants receiving anticoagulant therapy
* History of nasal abnormality (nasal surgery, trauma, polyp, obstruction)
* History of repeated epistaxis
* History of uncontrolled hypertension, diabetes, pregnancy, and any other cardiac or cerebral events.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Nasal bleeding | At the time of Intubation and Extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Mohtarma Benazir Bhutto Institute of Trauma, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient Confidentialit: Sharing IPD could compromise patient confidentiality and anonymity.
  Informed consent: Participants are not providing informed consent for their data to be shared and it could raise ethical concerns.

REFERENCES:
- [Background] Sato-Boku A, Sento Y, Kamimura Y, Kako E, Okuda M, Tachi N, Okumura Y, Hashimoto M, Hoshijima H, Suzuki F, Sobue K. Comparison of hemostatic effect and safety between epinephrine and tramazoline during nasotracheal intubation: a double-blind randomized trial. BMC Anesthesiol. 2021 Sep 30;21(1):235. doi: 10.1186/s12871-021-01454-y. PMID 34592949
- [Background] Ozkan ASM, Akbas S, Toy E, Durmus M. North Polar Tube Reduces the Risk of Epistaxis during Nasotracheal Intubation: A prospective, Randomized Clinical Trial. Curr Ther Res Clin Exp. 2018 Oct 9;90:21-26. doi: 10.1016/j.curtheres.2018.09.002. eCollection 2019. PMID 30787962
- [Background] Earle R, Shanahan E, Vaghadia H, Sawka A, Tang R. Epistaxis during nasotracheal intubation: a randomized trial of the Parker Flex-Tip nasal endotracheal tube with a posterior facing bevel versus a standard nasal RAE endotracheal tube. Can J Anaesth. 2017 Apr;64(4):370-375. doi: 10.1007/s12630-017-0813-4. Epub 2017 Jan 11. PMID 28078544
- [Background] Song J. A comparison of the effects of epinephrine and xylometazoline in decreasing nasal bleeding during nasotracheal intubation. J Dent Anesth Pain Med. 2017 Dec;17(4):281-287. doi: 10.17245/jdapm.2017.17.4.281. Epub 2017 Dec 28. PMID 29349350
- [Background] Patel S, Hazarika A, Agrawal P, Jain D, Panda NK. A prospective randomized trial of xylometazoline drops and epinephrine merocele nasal pack for reducing epistaxis during nasotracheal intubation. J Dent Anesth Pain Med. 2020 Aug;20(4):223-231. doi: 10.17245/jdapm.2020.20.4.223. Epub 2020 Aug 27. PMID 32934988